CLINICAL TRIAL: NCT04068714
Title: Retrospective Cohort Study of Open Versus Endovascular Repair of Abdominal Aortic Aneurysms
Brief Title: Open Versus Endovascular Repair of Abdominal Aortic Aneurysms
Status: Completed | Type: Observational
Sponsor: Hospital Sao Joao (Other)
Responsible Party: Principal Investigator, Marina Felicidade Dias Neto, Principal Investigator, Hospital Sao Joao
Other Study IDs: AAArepair
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Abdominal Aortic Aneurysm Without Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Endovascular repair: Observational retrospective cohort of patients consecutively submitted to elective abdominal aortic aneurysm surgery repair at a tertiary academic referral center from south Europe, between January 2009 and December 2015 through endovascular repair. The exclusion criteria were non-elective cases, aortic intervention due to diagnosis other than infrarenal AAA and complex aortic aneurysms such as juxta-renal, thoraco-abdominal or thoracic aneurysms.
  Interventions: Procedure: Type of aneurysm repair
- Open repair: Observational retrospective cohort of patients consecutively submitted to elective abdominal aortic aneurysm surgery repair at a tertiary academic referral center from south Europe, between January 2009 and December 2015 through open repair. The exclusion criteria were non-elective cases, aortic intervention due to diagnosis other than infrarenal AAA and complex aortic aneurysms such as juxta-renal, thoraco-abdominal or thoracic aneurysms.
  Interventions: Procedure: Type of aneurysm repair

INTERVENTIONS:
Procedure: Type of aneurysm repair — In open surgery repair group, aneurysm repair was performed by open surgery including aortobifemoral bypass, aorto-bi-iliac bypass and tubular aortic bypass. In endovascular repair (EVAR group), aneurysm correction was performed by percutaneous approach, femoral cutdowns and aorto-uni-iliac EVARs with femorofemoral bypass.

SUMMARY:
This is an observational retrospective cohort study of all patients consecutively submitted to elective abdominal aortic aneurysm surgery repair at a tertiary referral centre between 2009 and 2015. Patients were excluded if they were non-elective cases or had complex aortic aneurysms (juxta-renal, thoraco-abdominal or thoracic). Differences between both groups of repair were assessed, as well as short- and long-term complications including medical complications, duration of hospital stay, major cardiovascular events, mortality and vascular reintervention.

ELIGIBILITY:
Inclusion Criteria:

* This is an observational retrospective cohort study of all patients consecutively submitted to elective AAA surgery repair at a tertiary academic referral center from south Europe, between January 2009 and December 2015.

Exclusion Criteria:

* The exclusion criteria were non-elective cases, aortic intervention due to diagnosis other than infrarenal AAA and complex aortic aneurysms such as juxta-renal, thoraco-abdominal or thoracic aneurysms.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is an observational retrospective cohort study of all patients consecutively submitted to elective AAA surgery repair at a tertiary academic referral center from south Europe, between January 2009 and December 2015. The exclusion criteria were non-elective cases, aortic intervention due to diagnosis other than infrarenal AAA and complex aortic aneurysms such as juxta-renal, thoraco-abdominal or thoracic aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 12 months
  Acute myocardial infarction (with PCI, CABG or no intervention), decompensated heart failure, neurological deficit (including transient ischemic attack or stroke) or death

SECONDARY OUTCOMES:
Death | 12 months
  Death of any cause
Medical complications | 30 days
  Including digestive complications such as intestinal obstruction or ischemia, acute myocardial infarction (with PCI, CABG or no intervention), decompensated heart failure, neurological deficit (including transient ischemic attack or stroke), respiratory failure (including pneumonia, prolongation of endotracheal intubation, need for a tracheostomy) or acute renal failure (plasma creatinine > 3 mg/dL with or without the need for dialysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Universitário de São João, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No